CLINICAL TRIAL: NCT04768127
Title: ACHT - Adipositas Care & Health Therapy Zur Strukturierten, sektorenübergreifenden Versorgung Nach Bariatrisch-metabolischer Operation
Brief Title: Adipositas Care & Health Therapy
Acronym: ACHT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Deutsche Stiftung für chronisch Kranke (Unknown); Deutschen Gesellschaft für Allgemein- und Viszeralchirurgie e.V. (DGAV) (Unknown); AOK Bayern (Industry); Kassenärztliche Vereinigung Bayern (Unknown); symeda GmbH (Unknown); AMC Wolfartklinik Gräfelfing (Unknown); Schön Klinik Nürnberg Fürth (Unknown); Dr. Lubos Kliniken Bogenhausen (Unknown); Klinikum Memmingen (Unknown); Klinikum Passau (Unknown); Klinikum Nürnberg (Other); Helmholtz Zentrum München (Industry)
Responsible Party: Principal Investigator, Martin Fassnacht, Prof. Dr. Martin Fassnacht (Head of Endocrinolgy), Wuerzburg University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ACHT
Record Dates: First submitted 2020-12-16; First posted 2021-02-24 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Patients After Metabolic-bariatric Surgery; Obesity, Morbid
Keywords: bariatric surgery; patient adherence; post surgery care; morbid obesity; obesity surgery; obesity guide; aftercare program; electronic case file; obesity app; weight loss surgery
MeSH Terms: conditions — Obesity, Morbid; Patient Compliance

STUDY DESIGN:
Intervention Model Description: The study will compare two intervention groups (early intervention and later intervention) to two control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early aftercare (intervention group 1) (Experimental): Patients in this group will begin the ACHT program immediately after their bariatric metabolic operation. 3 weeks post surgery, they will attend the initial examination and meet their case manager. The obesity guide will then set up an electronic case file for the patient and introduce the patient to the obesity app. Through the next 18 months the obesity guide will monitor the patient's therapeutic success and adherence to the therapeutic goals. In month 2 patients visit a sports physician who assesses their mobility and physical capacity to compile a personal training plan, which will be uploaded onto the patient's case file and thus be available to the patient via the app. In months 3,6,9.12 and 18, patients will attend their aftercare appointments at specially trained ACHT physicians, where they will be physically examined by a physician and receive tailored dietary advice from a nutritional advisor. In month 18 patients revisit the surgical centre for the follow-up examination
  Interventions: Other: early aftercare
- Mid-term to long-term aftercare (intervention group 2) (Experimental): Patients in this group first visit the study center 18 months after their bariatric surgery for the initial examination and start the program in month 19 post-op. At the center, they will meet their obesity guide who will set up an electronic case file for the patient and introduce the patient to the obesity app. Throughout the next 18 months, the obesity guide will monitor the patient's therapeutic success and adherence to the therapeutic goals. In month 19 post-surgery, patients visit a sports physician who assesses their mobility and devises a personal training plan. This plan will be uploaded onto the patient's case file and made available to the patient via the app. In months 19,21,24, 30 and 36, patients attend their aftercare appointments at specially trained ACHT physicians, where they will be physically examined and receive tailored dietary advice. In month 36, patients will be reexamined at the study center.
  Interventions: Other: mid-term to late aftercare
- control group 1 (early aftercare) (No Intervention): Analogous to intervention group I, patients in this group are invited to the study center after verbal and written information. These patients will attend the one-off evaluation examination (18 months after the operation) at the obesity centre.
  If interested, patients in this group can be included in intervention group II until the required number of cases (140 patients) has been reached.
- control group 2 (mid-term to long-term aftercare) (No Intervention): Analogous to intervention group II, patients in this group are invited to the study center after verbal and written information. These patients will attend the one-off evaluation examination at the study center 36 months after the operation.

INTERVENTIONS:
Other: early aftercare — This group begins the aftercare program immediately after their bariatric surgery.
  Arms: Early aftercare (intervention group 1)
Other: mid-term to late aftercare — This group begins the aftercare program 18 months post surgery.
  Arms: Mid-term to long-term aftercare (intervention group 2)

SUMMARY:
ACHT - Adipositas Care and Health Therapy - is a structured, digitally-supported, cross-sectoral and close to home program developed for the postoperative care of patients following obesity surgery. The aim is to ensure the long-term success of therapy following bariatric surgery. ACHT was selected by the Federal Joint Commission for support under the Innovation Fund. The project started in July 2019 and will end in December 2022.

DETAILED DESCRIPTION:
In Germany, every second adult is overweight and almost one in four is obese - the trend is rising. Obesity is a chronic illness which significantly increases the risk of developing co-morbidities such as cardiovascular and joint diseases, cancer and diabetes. In addition to those functional and health limitations, many people are stigmatised which can lead to social exclusion and a reduced quality of life. Available conservative therapies do not always lead to sufficient, long-term weight loss. In those cases and if the disease is very pronounced, an obesity surgery (bariatric-metabolic surgery) can help. In order to ensure its success, patients require long-term after care following surgery. Currently, there are no necessary outpatient care standards and provisions. Inpatient obesity centres try to compensate for this with their own structures and limited resources, but are already reaching their limits.

The aim of the ACHT project is to ensure long-term therapeutic success after an operation. This is done through a digitally supported, structured, cross-sectoral and close-to-home aftercare program. Obesity case managers (obesity guides) coordinate the aftercare process and monitor the therapy goals. A digital case file links patients, case managers, resident doctors and obesity centers. Individual exercise goals, nutritional advice and psychological support are part of ACHT. ACHT is connected to quality assurance measures of a medical society.

Four groups are compared in the ACHT study. One group begins their 18 months ACHT aftercare program directly after the operation, another group 18 months after the operation. These two groups are compared to patients who receive standard care. Through these two intervention groups, we hope to examine the long-term effects of the program within the given time constraints of the study.

ACHT is funded for three and a half years by the Federal Joint Committee as part of the Innovation Fund with approx. 4.5 million euros.

ELIGIBILITY:
Inclusion Criteria:

relevant for all groups:

* patients who have already approved to have their data entered into the National Registry of metabolic and bariatric diseases (StuDoQ, DGAV)
* Sufficient knowledge of the German language to use the app, to communicate with the obesity case manager (obesity guide) and to fill out the questionnaires
* signed consent form

group specific criteria:

Intervention group I ("early aftercare"):

* Insured with the Allgemeine Ortskrankenkasse (AOK) Bayern
* Consent to participate in the selective contract
* The bariatric metabolic operation (sleeve gastrectomy, Roux-en-Y-gastric bypass) was carried out 3 weeks (+/- 10 days) before the entrance examination
* iOS or Android smartphone (operating system: iOS 11 or higher or Android 6 or higher) with internet access can be used for study
* Sufficient mobility to get to the aftercare practice regularly and to complete an exercise program

Intervention Group II ("medium-term and late after care") recruited from control group I:

* Insured with the Allgemeine Ortskrankenkasse (AOK) Bayern
* Consent to participate in the selective contract
* The bariatric-metabolic operation (sleeve gastrectomy or Roux-en-Y-gastric bypass) was carried out 18 months (+/- 2 months) before time of recruitment

Control group I (compared to early intervention):

* Insured with the Allgemeine Ortskrankenkasse (AOK) Bayern
* The bariatric metabolic operation was carried out 18 months (+/- 2 months) before time of recruitment
* Sufficient mobility (see intervention group, so that groups are comparable)

Control group II (compared to late intervention):

* The bariatric metabolic operation was carried out 36 months (+/- 2 months) before the recruitment date
* Sufficient mobility (see intervention group, so that groups are comparable)
* The health insurance is irrelevant in this group

Exclusion Criteria:

* State after a revision operation
* Planned two-stage surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified King's Score (comparison between intervention group I and control group I resp. intervention group II and control group II) | 18 months
  Primary endpoint will be the difference in the modified King's Score between intervention group I and control group I resp. intervention group II and control group II. The modified King's Score is a multifaceted sum score taking into account categories A to L (airways, BMI, cardiovascular, diabetes mellitus, economic, functional, gonadal/sexuality, health status, body image, junction (gastroesophageal), kidney, liver). For each category patients receive between 0 and 3 points describing the degree of impairment (0 Points: normal; 3 Points: severe impairment); the minimum score can be 0, maximum sum score can thus be 36.

SECONDARY OUTCOMES:
General Quality of life | 18 months
  Quality of life is measured by Short Form 36 (SF-36); Minimum 0 Points, Maximum 100 Points; higher values mean a better outcome
Bariatric Quality of life | 18 months
  Quality of life is measured by Bariatric Quality of life (BQL); Minimum 13 Points, Maximum 65 Points; higher values mean a better outcome
Health-specific Quality of life | 18 months
  Quality of life is measured by EuroQuol-5 dimensions (EQ-5D); each of the 5 dimensions has between 1 Point (no Limitation in that Dimension) and 5 Points (severe Limitation in that Dimension)
- Depression | 18 months
  Depression is measured by Patient Health Questionnaire 9 (PHQ-9 questionnaire); Minimum 0 Points, Maximum 27 Points, lower values mean better outcome
- Single dimensions of the modified King's Score | 18 months
  - Single dimensions of the modified King's Score
Percentage of Patients with folic acid deficiency | 18 months
  - Measurement of folic acid (ng/ml); percentage of patients with values below the reference range
Percentage of Patients with Vitamin B 12 deficiency | 18 months
  - Measurement of Vitamin B 12 (pg/ml); percentage of patients with values below the reference range
Percentage of Patients with Vitamin B 1 deficiency | 18 months
  - Measurement of Vitamin B 1 (µg/l); percentage of patients with values below the reference range
Percentage of Patients with Vitamin B 6 deficiency | 18 months
  - Measurement of Vitamin B 6 (µg/l); percentage of patients with values below the reference range
Percentage of Patients with iron deficiency | 18 months
  - Measurement of ferritin (µg/l); percentage of patients with values below the reference range
Percentage of Patients with protein deficiency | 18 months
  - Measurement of prealbumin (mg/dl); percentage of patients with values below the reference range
Percentage of patients with symptoms of postoperative malnutrition based on 9 standardized questions | 18 months
  - Postoperative nutritional status will be assessed via 9 questions from a standardized questionnaire (StuDoQ DGAV); questions can be answered by "yes" or "no"; number of questions answered by "yes"
Percentage of Procedure-specific long term complications: Dumping syndrome | 18 months
  percentage of patients with Dumping syndrome (Patients will be asked for symptoms)
Percentage of Procedure-specific long term complications: gastric ulcers | 18 months
  percentage of patients with gastric ulcers (Patients will be asked for symptoms and findings if endoscopy was performed)
Percentage of Procedure-specific long term complications: gall stones | 18 months
  percentage of patients with gall Stones (Patients will receive a sonography of the gall bladder)
Percentage of Procedure-specific long term complications: internal hernia | 18 months
  percentage of patients with internal hernia (Patients are asked if they had surgery for internal hernia)
percentage of procedure-specific long term complications: anastomosis Stenosis | 18 months
  percentage of Patients with anastomosis Stenosis (Patients will be asked for recurrent vomiting and if an endoscopic or surgical Intervention was performed)
Change in lean Body mass | 18 months
  - Body composition will be assessed by bioelectrical impedance Analysis measuring the percentage of lean Body mass
Change in Phase angle | 18 months
  - Body composition will be assessed by bioelectrical impedance Analysis measuring the Phase angle
average number of Sick days | 18 months
  Average number of Sick days in the past 12 months (information provided by the Patient and data of the respective health insurance)
- Patient adherence | 18 months
  number of attended appointments
Percentage of patients reaching their Goal for steps per day | 18 months
  Percentage of Patients achieving their treatment goal for steps per day, comparison between individual goal (defined according to the physical working capacity 120) and state at study inclusion
Percentage of patients reaching their Treatment Goal for physical activity | 18 months
  Percentage of Patients achieving their treatment goal for physical activity, comparison between individual goal (defined according to the physical working capacity 120) and state at study inclusion
- Acceptance of the ACHT aftercare program | 18 months
  - Acceptance of the ACHT aftercare program by patients and professionals (physicians, nutritionists) measured by a self-designed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Zippel-Schultz, PhD, Study Director — Deutsche Stiftung für chronisch Kranke; Martin Fassnacht, MD, Principal Investigator — Wuerzburg University Hospital
Locations (7):
- Germany (7):
  - AMC WolfartKlinik, Zentrum für Adipositas- und Metabolische Chirurgie, Gräfelfing
  - Adipositaszentrum Klinikum Memmingen, Memmingen
  - Chirurgische Klinik München-Bogenhausen GmbH, München
  - Klinikum Nürberg, Nuremberg
  - Sana Klinikum Offenbach GmbH, Offenbach
  - Klinikum Passau, Passau
  - Wuerzburg University Hospital, Würzburg